CLINICAL TRIAL: NCT07246200
Title: Evaluation of Standard TED Stocking vs. Reparel Bioactive Garment on Postoperative Leg Swelling, Pain and DVT Rates After Hip Replacement Surgery
Brief Title: TED Stocking vs. Reparel Garment After Hip Replacement
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Reparel (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 111225
Record Dates: First submitted 2025-11-13; First posted 2025-11-24 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Osteoarthritis (OA) of the Hip
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Bioactive Sleeve on Operative Leg (Experimental): Participants receive the Reparel Bioactive Sleeve on the operative leg and the Standard TED Stocking on the non-operative leg.
  Interventions: Device: Reparel Bioactive Sleeve
- Bioactive Sleeve on Non-Operative Leg (Active Comparator): Participants receive the Reparel Bioactive Sleeve on the non-operative leg and the Standard TED Stocking on the operative leg.
  Interventions: Device: TED Stocking

INTERVENTIONS:
Device: Reparel Bioactive Sleeve — A non-compressive, photobiomodulating sleeve worn on the leg to reduce postoperative pain and swelling.
  Arms: Bioactive Sleeve on Operative Leg
Device: TED Stocking — Standard-of-care gradient compression stocking used after hip replacement.
  Arms: Bioactive Sleeve on Non-Operative Leg

SUMMARY:
This randomized, prospective study compares the effectiveness of a novel bioactive garment (Reparel Leg Sleeve) versus standard TED compression stockings in reducing postoperative leg swelling, pain, and deep vein thrombosis (DVT) rates following total hip arthroplasty. The study aims to determine whether the bioactive garment improves patient comfort and recovery outcomes compared to traditional stockings.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-89
* Undergoing primary unilateral total hip replacement
* BMI < 40
* Able to follow postoperative protocol
* English speaking

Exclusion Criteria:

* Age <18 or >90
* Physical inability to use stockings
* Allergy to silicone/polyester
* Active DVT
* History of vascular bypass on operative limb (e.g., Fem-Pop, Fem-Fem)
* Inability to comply with post-op/rehab
* Lymphedema

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2024-01-01 (Actual); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Pain Score (VAS) | Postoperative Weeks 2, 6, and 12
  Pain will be measured using the Visual Analog Scale (VAS), a standard 0-10 numeric rating scale. Patients will report pain levels during routine postoperative follow-up visits or via validated questionnaires.
HOOS Jr. Score | Postoperative Weeks 6 and 12
  The Hip Disability and Osteoarthritis Outcome Score, Junior (HOOS Jr.) evaluates hip function and patient-reported symptoms following total hip arthroplasty.
VR-12 Score | Postoperative Week 12
  The Veterans RAND 12-Item Health Survey (VR-12) evaluates patient-reported physical and mental health status.
HSS Satisfaction Score | Postoperative Week 12
  The Hospital for Special Surgery (HSS) Satisfaction Score assesses patient satisfaction following hip replacement surgery.
Forgotten Joint Score | Postoperative Week 12
  The Forgotten Joint Score measures the extent to which patients are aware of their hip joint during daily activities, reflecting functional recovery.

SECONDARY OUTCOMES:
Leg Swelling (Clinical Evaluation) | Postoperative Weeks 2, 6, and 12
  Leg swelling will be assessed during routine postoperative clinic visits through standard clinical evaluation, including circumferential measurement and visual assessment for edema.
Incidence of Deep Vein Thrombosis | Up to 12 weeks after surgery
  Deep vein thrombosis (DVT) occurrence will be monitored through standard postoperative care, including clinical evaluation and diagnostic testing if symptoms suggest DVT.
Postoperative Narcotic Use | Collected at 2, 6, and 12 weeks after surgery
  Self-reported narcotic medication use will be documented through postoperative questionnaires to compare pain-management differences between intervention assignments.
Study Questionnaire Responses | Weeks 2, 6, and 12 postoperatively
  Patients will complete a study-specific questionnaire assessing comfort, usability, perceived swelling, and overall satisfaction with the leg garments.

CONTACTS AND LOCATIONS:
Locations (1):
- Institute for Joint Restoration, Fremont, California, United States

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (2):
  • Study Protocol (2021-12-01): https://cdn.clinicaltrials.gov/large-docs/00/NCT07246200/Prot_000.pdf
  • Informed Consent Form (2023-01-20): https://cdn.clinicaltrials.gov/large-docs/00/NCT07246200/ICF_001.pdf